CLINICAL TRIAL: NCT03846934
Title: Positive and Quantitative Diagnosis of Pleural Effusions by Thoracic Ultrasonography in Patients With Acute Respiratory Failure in the Emergency Department
Acronym: POCUYTO
Status: Terminated | Type: Observational
Why Stopped: enough patients
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI18_032 (POCUYTO)
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Pleural Effusion; Ultrasonography; Thoracic; Acute Respiratory Failure; Emergencies
Keywords: Pleural Effusion; Ultrasonography; Thoracic; Acute Respiratory Failure; Emergencies
MeSH Terms: conditions — Pleural Effusion; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasonography thoracic: Ultrasonography thoracic
  Interventions: Device: Ultrasonography thoracic

INTERVENTIONS:
Device: Ultrasonography thoracic — Thoracic ultrasonography will be performed as soon as possible after admission to the ED, without delaying the start of treatment and in addition to routine thoracic radiography.

SUMMARY:
Acute respiratory failure (ARF) is a frequent reason for consulting in the Emergency Department (ED) and one of the major clinical problems prompting admission in intensive care unit. In the ED, evaluation of an ARF is mainly based on clinical examination and frontal chest x-ray performed to the patient bedside. This practice has a limited diagnostic capacity due to a lack of specificity of clinical and radiological semiology, especially in the polypathological patient. Thoracic ultrasonography provides morphological information regrouped as a syndrome (interstitial syndrome, alveolar condensation, pneumothorax) and allows the identification of pleural effusions (PE). The PE diagnosis is easy, quick, and relies on two-dimensional ultrasound imaging. Compared to CT scan, which remains the reference examination although ill-suited in the context of emergency, thoracic ultrasonography has a sensitivity and specificity greater than 90% for pleural liquid (PL) diagnosis. In addition, thoracic ultrasonography is used to assess the volume of PL, determine its nature and guide the pleural puncture with higher performance than chest x-ray. The semi-quantitative evaluation of PEs has been validated in patients with mechanical ventilation hospitalized in intensive care unit. On the other hand, few data on the prevalence and quantification of PL for hospitalized patients in ED for an ARF are currently available.

Thus, the objective of this study is to evaluate the prevalence and severity of the PL identified by thoracic ultrasonography in patients admitted to the ED for an ARF by emergency physicians with ultrasound skills recommended by the French Society of Emergency Medicine.

DETAILED DESCRIPTION:
Acute respiratory failure (ARF) is a frequent reason for consulting in the Emergency Department (ED) and one of the major clinical problems prompting admission in intensive care unit. In the ED, evaluation of an ARF is mainly based on clinical examination and frontal chest x-ray performed to the patient bedside. This practice has a limited diagnostic capacity due to a lack of specificity of clinical and radiological semiology, especially in the polypathological patient. Thoracic ultrasonography provides morphological information regrouped as a syndrome (interstitial syndrome, alveolar condensation, pneumothorax) and allows the identification of pleural effusions (PE). The PE diagnosis is easy, quick, and relies on two-dimensional ultrasound imaging. Compared to CT scan, which remains the reference examination although ill-suited in the context of emergency, thoracic ultrasonography has a sensitivity and specificity greater than 90% for PL diagnosis. In addition, thoracic ultrasonography is used to assess the volume of PL, determine its nature and guide the pleural puncture with higher performance than chest x-ray. The semi-quantitative evaluation of PEs has been validated in patients with mechanical ventilation hospitalized in intensive care unit. On the other hand, few data on the prevalence and quantification of PL for hospitalized patients in ED for an ARF are currently available.

Thus, the objective of this study is to evaluate the prevalence and severity of the PL identified by thoracic ultrasonography in patients admitted to the ED for an ARF by emergency physicians with ultrasound skills recommended by the French Society of Emergency Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the ED
* AND Age >= 18 years
* AND affiliated or beneficiary to a social security scheme
* AND with clinical signs of ARF:

  * Cyanosis, mottling, encephalopathy
  * Respiratory exhaustion (thoraco abdominal balancing, accessory muscle play)
  * Pulse oxygen saturation (SpO2) <92% in the air
* AND/OR showing biological signs of ARF:

  * Arterial oxygen pressure (PaO2) <60 mmHg
  * Or PaO2 / fraction of inspired oxygen (FiO2) ratio <400.

Exclusion Criteria:

* Patient moribund or for whom a limitation of the care is envisaged
* Pregnant woman
* Absence of exploitable ultrasound image for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted to ED and presenting with clinical signs of ARF
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Clinically relevant Pleural Effusions (PE) | Day 1
  Number and proportion of ARF patients for whom the thoracic ultrasonography realized in ED shows a clinically relevant PE (> 2cm)

SECONDARY OUTCOMES:
Inter-pleural distance to the inspiration | Day 1
  Measuring of the inter-pleural distance to the inspiration (patient in spontaneous ventilation) in cross-section
Additional diagnostic elements | Day 1
  Number and proportion of patients for whom the thoracic ultrasound provides additional diagnostic evidence in comparison to clinical examination and the standard thoracic radiography in frontal bed, ie:
  Presence of an PE Abundant PE> 800 mL Or any other pleuro-parenchymal abnormalities identified by ultrasound (pneumothorax, condensation of lung parenchyma ...) and not on standard radiography

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No